CLINICAL TRIAL: NCT04440527
Title: Intraocular Pressure After Preserflo /Innfocus Microshunt vs Trabeculectomy: a Prospective, Randomised Control-trial (PAINT-Study)
Brief Title: Intraocular Pressure After Preserflo / Innfocus Microshunt Implantation vs Trabeculectomy
Acronym: PAINT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PAINT-Study
Record Dates: First submitted 2020-06-18; First posted 2020-06-19 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Primary Open Angle Glaucoma; Pseudoexfoliation Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Exfoliation Syndrome | interventions — Trabeculectomy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microshunt (Experimental): Patients will be treated with Preserflo / Innfocus Microshunt (Santen Pharmaceutical Co., Ltd.).
  Interventions: Device: Preserflo / Innfocus Microshunt
- Trabeculectomy (Active Comparator): Patients will be treated with trabeculectomy.
  Interventions: Other: Trabeculectomy

INTERVENTIONS:
Device: Preserflo / Innfocus Microshunt — The Microshunt features an 8.5-mm tube with an outer diameter of 350 µm and a 70-µm diameter lumen. Implantation creates a subconjunctival bleb and lowers intraocular pressure by increasing aqueous humor outflow.
  Arms: Microshunt
Other: Trabeculectomy — Trabeculectomy is the most commonly performed surgical procedure and is considered the gold standard.
  Arms: Trabeculectomy

SUMMARY:
The aim of this project is to compare trabeculectomy with Preserflo / Innfocus Microshunt in patients with Primary Angle Open Glaucoma and Pseudoexfoliation Glaucoma regarding the reduction of intraocular pressure.

DETAILED DESCRIPTION:
The study is a prospective, randomized, monocentric, part blinded, controlled non-inferiority study of glaucoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Primary open angle glaucoma or pseudoexfoliation glaucoma
* medically uncontrollable intraocular pressure or intolerance of topical therapy
* negative urine/serum pregnancy test of women in childbearing age
* signed and dated informed consent

Exclusion Criteria:

* previous incisional glaucoma procedure on affected eye
* pregnancy, nursing period
* Patients in military service, training periods and civil service
* Participation in another clinical trail
* pre-existing ocular pathologies: high myopia (refraction ≥8.00 D), thin conjunctiva

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-07-22 (Estimated); Primary Completion 2022-07-22 (Estimated); Study Completion 2024-07-22 (Estimated)

PRIMARY OUTCOMES:
Difference in intraocular pressure | 1 year
  The primary endpoint is the difference between intraocular pressure after microshunt implantation vs trabeculectomy.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: Undecided